CLINICAL TRIAL: NCT05709912
Title: Randomized Controlled Trial of a Psychosocial Mobile Application (App) to Promote Coping for Caregivers of Patients Receiving Hematopoietic Cell Transplantation (HCT)
Brief Title: Mobile CARE-App to Promote Coping for Caregivers of Patients Receiving Stem Cell Transplant
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-634
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Bone Marrow Transplant Complications; Hematologic Malignancy
Keywords: Cognitive Behavioral Therapy; CBT; Hematopoietic stem cell transplantation; HCT; Bone Marrow Transplant Complications; Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARE App (Experimental): Participants randomized to the CARE app + usual care will complete the following:
  * Questionnaires at baseline, Day 10, Day 60, and Day 100 post-HCT
  * use the CARE app from enrollment up to 60 days post-HCT: the CARE app includes 5 contains 5 modules and a 6th optional module
  * receive usual care as per HCT practice which entails meeting with a transplant social worker prior to HCT and as needed for extra visits
  Interventions: Behavioral: CARE Application
- Usual Care (Active Comparator): Participants randomized to usual care will complete the following:
  * Questionnaires at baseline, Day 10, Day 60, and Day 100.
  * receive usual care as per HCT practice, which entails meeting with a transplant social worker prior to HCT and as needed for extra visits.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: CARE Application — Self-administered, psychosocial mobile application comprised of 5 learning modules.
  Arms: CARE App
Behavioral: Usual Care — Meeting with transplant social worker prior to HCT, consistent with standard-of-care.
  Arms: Usual Care

SUMMARY:
The goal of this research study is to determine whether a self-administered, psychosocial mobile application (CARE app) is effective at improving the quality of life and experience of caregivers of patients receiving hematopoietic stem cell transplantation (HCT).

DETAILED DESCRIPTION:
This is a randomized clinical trial to determine whether a psychosocial mobile application (CARE app) is effective at improving the quality of life and experience of caregivers of patients receiving hematopoietic stem cell transplantation (HCT). The CARE app was developed with the goal of addressing the needs of caregivers of HCT recipients.

Participants will be randomized into one of two study groups: CARE app plus Usual Care versus Usual Care.

Participation in this study is expected to last up to 100 days after HCT.

It is expected that about 120 people will take part in this research study.

The Leukemia and Lymphoma Society is supporting this research by providing funding.

ELIGIBILITY:
Caregiver Inclusion Criteria:

* Adult caregivers (>18 years) who is a relative or friend who live with the patient or is a designated caregiver as indicated during the transplant process.
* Caregiver of a patient receiving allogeneic or autologous HCT for the treatment of cancer
* Ability to comprehend and speak English as the CARE app is only available in English

Patient Exclusion Criteria:

* Caregivers of patients undergoing HCT for benign hematologic conditions
* Caregivers with acute or unstable psychiatric or cognitive conditions which the treating clinicians believes prohibits informed consent or compliance with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Caregiver quality of life (QOL) as measured by the Caregiver Oncology Quality of Life (CARGOQOL) questionnaire | up to 60 days post-HCT
  Compare caregiver QOL as measured by the CARGOQOL between the two study groups. The CARGOQOL ranges from 0-100 with higher scores indicating better QOL

SECONDARY OUTCOMES:
Caregiver quality of life (QOL) as measured by the Caregiver Oncology Quality of Life (CARGOQOL) questionnaire | up to 100 days post HCT
  Compare caregiver QOL as measured by the CARGOQOL between the two study groups longitudinally. The CARGOQOL ranges from 0-100 with higher scores indicating better QOL
Caregiving burden as measured by the Caregiver Reaction Assessment (CRA) | Up to 100 days post HCT
  Compare caregiving burden as measured by the CRA between the two study groups. The CRA ranges from 24-120 with higher scores indicating greater caregiving burden
Anxiety symptoms as measured by the Hospital Anxiety and Depression scale (HADS-Anxiety) | Up to 100 days post HCT
  Compare anxiety symptoms as measured by the HADS-Anxiety between the study groups. The HADS-Anxiety ranges from 0-21 with higher scores indicating worse anxiety symptoms
Depression symptoms as measured by the Hospital Anxiety and Depression Scale (HADS-Depression) | Up to 100 days post HCT
  Compare depression symptoms as measured by the HADS-Depression between the study groups. The HADS-Depression ranges from 0-21 with higher scores indicating worse depression symptoms
Post-traumatic stress symptoms (PTSD) as measured by the PTSD Checklist | Up to 100 days post HCT
  Compare post-traumatic stress symptoms as measured by the Post-Traumatic Stress Checklist-Civilian Version between the two groups. The checklist ranges from 17-85 with higher scores indicating worse PTSD Symptoms

OTHER OUTCOMES:
Coping as measured by the Measure of Current Status (MOCS) | Up to 100 days post-HCT
  Comparing caregiver coping as measured by the MOCS between the two study groups. The scale ranges from 0-52 with higher scores indicating higher coping skills
Self-efficacy as measured by the Cancer self-efficacy-transplant (CASE-t) scale | Up to 100 days post-HCT
  Compare caregiver self-efficacy as measured by the CASE-t between the two study groups. The scale ranges from 0-170 with higher scores indicating better self-efficacy
Usability of the CARE app using the System Usability Scale | up to 60 days post-HCT
  Assess the usability of the care app (in those receiving the intervention) using the System Usability Scale, which ranges 0-100 with higher scores indicating better usability

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Willis KD, Barata A, Freese M, Applebaum AJ, Nelson A, Traeger LN, Horick NK, Rabideau DJ, Temel JS, Greer JA, Jacobs JM, El-Jawahri A. Randomised controlled trial of a psychosocial digital health application to promote coping for caregivers of patients undergoing haematopoietic stem cell transplantation: a study protocol for the BMT-CARE app. BMJ Open. 2025 Apr 8;15(4):e092371. doi: 10.1136/bmjopen-2024-092371. PMID 40204300